CLINICAL TRIAL: NCT01043848
Title: Therapeutic Effects of Early and Late Onset Peripheral Pudendal Neurostimulation on Bladder Function and Autonomic Neuroplasticity in SCI - a Controlled European Multicenter Study
Brief Title: Treatment of Neurogenic Detrusor Overactivity: Early Versus Late Pudendal Nerve Stimulation in Spinal Cord Injury (SCI) Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient recruitment, necessary number of patients could not be included within the required time frame
Sponsor: Ulrich Mehnert (Other)
Collaborators: Institut Guttmann (Other); Schweizerisches Paraplegikerzentrum Nottwil (Unknown); BG Unfallklinik Murnau (Other); Klinik für Paraplegiologie, Universitätsklinikum Heidelberg (Unknown)
Responsible Party: Sponsor-Investigator, Ulrich Mehnert, Executive physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMSCI-NU-2/09
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Neurogenic Detrusor Overactivity; Spinal Cord Injury
Keywords: neurogenic detrusor overactivity; neuromodulation; spinal cord injury; pudendal nerve stimulation; videocystometry; neurophysiology; neuroplasticity
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (3):
- Early pudendal stimulation (Experimental): Subjects in this arm will start with the intervention within 2 weeks after SCI
  Interventions: Procedure: external electric pudendal nerve stimulation
- Late pudendal stimulation (Experimental): Subjects in this arm will start with the intervention 12 weeks after SCI
  Interventions: Procedure: external electric pudendal nerve stimulation
- Control (No Intervention): Subjects in this arm will be treated according to standard therapy but will receive no pudendal stimulation

INTERVENTIONS:
Procedure: external electric pudendal nerve stimulation — intervention timing: twice daily for 20 minutes during 3 consecutive months.
  intervention procedure: electrodes will be placed around the penile shaft (in males) or clips will be directly placed on the clitoris (in females).
  intervention device: contic+
  stimulation parameters: 10 Hz, 200μs pulse width, 10mA (or less, if too uncomfortable).
  Other Names: contic+, tic Medizintechnik GmbH, 46286 Dorsten, Germany
  Arms: Early pudendal stimulation; Late pudendal stimulation

SUMMARY:
Background: Although a small group, special attention has to be given to lower urinary tract (LUT) dysfunctions in spinal cord injury (SCI) patients, as they also suffer under a loss of motor-sensory function and autonomic regulation next to the severe deficiencies in bladder and bowel control. Autonomic dysregulation linked with LUT dysfunction can cause autonomic dysreflexia with life threatening increases in blood pressure and there is still no concept for an early rehabilitation of bladder function after SCI.

Hypothesis: We assume that inadequate reorganization of nerve fibres in SCI is a reason for spastic bladder dysfunction and vegetative dysregulation and that this can be positively influenced by early neuromodulation. We hypothesized that bladder dysfunction as well as autonomic dysreflexia will be positively affected.

Specific aims: Evaluation, if external pudendal nerve stimulation (EPS) can positively influence LUT rehabilitation in SCI patients and if early initiation of stimulation is more effective compared to late initiation (after spinal shock).

Experimental design: Prospective multicentre study in 36 SCI patients (24 treatment subjects, 12 control subjects). EPS will be started either within 10 days after SCI (early stim group) or after cessation of spinal shock (late stim group). Effects on spastic bladder function and autonomic disinhibition will be assessed by urodynamics, vegetative tests, and by electrophysiological techniques.

Expected value: If early EPS is effective and complete SCI patients benefit from this intervention; and if early onset of EPS has better and longer lasting effects than late onset stimulation, the findings will be of utmost relevance not only for bladder function but also to alleviate adverse phenomena such as autonomic dysreflexia. Neurostimulation may bear the opportunity to early reshape maladaptive neuroplasticity. This would be proof of an effective modulation and promotion of neuroplasticity, thus opening up new treatment options in the field of paraplegiology.

ELIGIBILITY:
Inclusion Criteria:

* Single event traumatic or ischemic Para- or Tetraplegia
* Complete SCI (ASIA A)
* Lesion level between C4 and Th10
* Performance of study treatment and assessments possible according to the study time schedule
* Patient capable and willing of giving written informed consent

Exclusion Criteria:

* Nontraumatic Para- or Tetraplegia (i.e. disc herniation, tumor, AV- Malformation, myelitis) exkl. single event ischemic incidences
* Pre- known dementia or severe reduction of intelligence, leading to reduced capabilities of cooperation or giving consent
* Peripheral Nerve lesions below the level of lesion (i.e. pudendal nerve impairment, cauda equina syndrome, pre- known Polyneuropathy)
* Severe craniocerebral injury
* Previous or planned intradetrusor injections of botulinum toxin
* Previous or planned surgical therapy for neurogenic detrusor overactivity (e.g. bladder augmentation, Mitrofanoff, sphincter prothesis, sacral neuromodulation, deafferentation, sphincterotomy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Videocystometry | week 4, 12, 26, 38, 52 after SCI

SECONDARY OUTCOMES:
Neurophysiological measurements (NCV, BCR, SSR) | week 2, 4, 12, 26, 38, 52 after SCI

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mehnert, MD, Principal Investigator — University of Zurich; Martin Schubert, MD, Principal Investigator — Balgrist University Hospital
Locations (3):
- Guttmann Institute, Badalona, Barcelona, Spain
- Switzerland (2):
  - Schweizerisches Paraplegikerzentrum Nottwil, Nottwil, Canton of Lucerne
  - Balgrist University Hospital, Zurich